CLINICAL TRIAL: NCT00524823
Title: Early Detection of Prostate Cancer by FACS
Acronym: FACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Other Study IDs: HP 7-251 S
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-08

CONDITIONS: Prostate Cancer; Hyperplasia
Keywords: Prostate Cancer; Hyperplasia - BPH; FACS; Prostate Cancer, Hyperplasia - BPH, Malignancy
MeSH Terms: conditions — Prostatic Neoplasms; Hyperplasia; Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: 10 diagnosed men in age 60 - 90 with Prostate Cancer
- 2: 10 patients with benign growth
- 3: 10 health volunteers
- 4: 10 patients diagnosed with other cancer

SUMMARY:
Early detection of prostrate cancer and development of metastases. The research will attempt to match the SCM test (structuredness of the cytoplasmic matrix) in lymphocytes as an early cancer detection test using Florescent Activated Cell Sorting (FACS) as a replacement for the CellScan instrument. The test is based on measurement of cellular changes in response to the specific prostate antigen, PSA.

ELIGIBILITY:
Inclusion Criteria:

Experimental group : Males between the ages of 60-90 years, with medical diagnosis of prostate cancer according to both clinical and hematological examinations, before receiving any medical treatment.

Control Group 1: Males between the ages of 60-90 years, with diagnosed benign prostate hyperplasia -BPH.

Control Group 2: Males between the ages of 60-90 years, medically diagnosed as healthy.

Control Group 3: Males between the ages of 60-90 years, medically diagnosed with another form of cancer, not prostate.

Exclusion Criteria:

Experimental group: Other known cancer or systemic infection. Control Group 1: Other known cancer or systemic infection. Control Group 2:Past hematological disorders nor cancer growth history. other known systemic infection, nor urinary tract infection. Patients hospitalized for orthopedic injuries of any type who are otherwise free of urinary tract infections.

Control Group 3:Other known systemic infection, nor urinary tract infection.

-

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kucherski, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Urology Department, Ziv Medical Center, Safed, Israel

REFERENCES:
- [Background] Klein O, Lin S, Embon O, Sazbon A, Zidan J, Kook AI. An approach for high sensitivity detection of prostate cancer by analysis of changes in structuredness of the cytoplasmic matrix of lymphocytes specifically induced by PSA-ACT. J Urol. 1999 Jun;161(6):1994-6. PMID 10332488
- [Background] Altman, Roberta. The prostate Answer Book. Warner Books, lnc., 1993.
- [Background] American Cancer Society. National Cnference on Prostate Cancer. Philadelphia, Pennsylvania: September/October 1994.
- [Background] Rous, Stephen N., M.D.; The prostate Book. W.W. Norton & Co., 1992.